CLINICAL TRIAL: NCT00001468
Title: Outcomes of Education and Counseling for BRCA1 or BRCA2 Testing
Brief Title: Outcomes of Education and Counseling for BRCA1 Testing
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950085; 95-HG-0085
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Breast Neoplasms; Ovarian Neoplasms
Keywords: Behavioral and Attitudinal Changes; Breast Cancer; High Risk Families; Inherited Susceptibility; Psychological Responses to Risk
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Behavior; Genetic Predisposition to Disease

SUMMARY:
This study will identify how personal beliefs, values and family experiences affect a person's decision as to whether or not to be tested for changes in a gene called BRCA1 or BRCA2. Changes in these genes are associated with a significantly increased risk of breast and ovarian cancer in women, a slightly higher risk of prostate cancer in men, and a slightly higher risk of colon cancer in both men and women.

Families enrolled in the National Cancer Institute's familial cancer research project who also participated in a telephone survey (protocol 78-C-0039) regarding their level of interest in BRCA1/2 testing results may be eligible for this study.

All participants will complete a 20- to 30-minute questionnaire assessing knowledge, risk perception and personality traits, and will participate in an education session to review the following:

* Information about their individual cancer risk, based on family history
* Potential benefits and risks (medical, psychological and social) of BRCA1/2 testing, both for those who test positive and those who test negative
* Overview of DNA testing (what is done and how accurate it may or may not be)
* Medical management options for those at increased risk for breast and ovarian cancer
* Environmental cancer risk factors
* Instruction in breast self-examination

Participants will then be asked whether or not they want to undergo BRCA1/2 testing

Those who want to be tested will be divided into two groups to compare counseling methods (client-centered vs. counselor-driven counseling). A small blood sample (2 to 3 tablespoons) will be drawn for genetic analysis. Test results will be provided in person at a second visit-this may take 6 months or more. A follow-up telephone call 2 weeks after receipt of the test results will address participants' questions and provide support. During a third visit, scheduled 6 months after receipt of the test results, participants will complete questionnaires evaluating mood, attitude, self-esteem, family interactions, cancer screening practices, and other factors. Finally, 1 year after receipt of the test results, participants will be contacted by telephone and asked about their feelings about the test and its outcome.

Individuals who choose not to have gene testing will not participate in any in-person sessions after the initial visit. They will be followed with no more than two telephone interviews to assess their feelings and attitudes related to their decision not to be tested.

Individuals may reconsider and change their mind at any time regarding their decision-whether to be tested or not.

The results of the study will help experts devise the most effective methods of educating and counseling people at high risk for having an altered BRCA1/2 gene.

DETAILED DESCRIPTION:
Women at increased risk for developing breast and/or ovarian cancer and their first degree relatives will be offered BRCA1/2 gene testing. This study proposes to evaluate psychological and behavioral aspects of their decision-making and the outcomes of the testing process. Knowledge and expectations will be assessed initially, followed by pre-test psychological assessment and an in person education and counseling session. Participants will be presented the choice of whether or not to undergo BRCA1/2 testing. Notification of test results will occur in person along with discussion of available surveillance options. Telephone interviews will assess psychological and behavioral outcome measures at 6 and/or twelve month time points. Aspects of this research endeavor have been designed to complement an NHGRI/NCI extramural consortium and an NHGRI/NCI intramural collaboration both of which will address various aspects of risk notification and follow-up for hereditary breast, ovarian and colon cancer.

ELIGIBILITY:
Participants will be drawn from the families enrolled by Drs. Peggy Tucker and Jeff Struewing in the GEB of NCI (protocol 78-C-0039).

Individual with a family history of verified breast and/or ovarian cancer that includes;

1. two cases of ovarian cancer in first degree relatives, or
2. three cases of breast cancer and at least one case of ovarian cancer (two of which have to be first degree relatives), or
3. at least four cases of breast cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 1995-03; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Biesecker BB, Boehnke M, Calzone K, Markel DS, Garber JE, Collins FS, Weber BL. Genetic counseling for families with inherited susceptibility to breast and ovarian cancer. JAMA. 1993 Apr 21;269(15):1970-4. PMID 8352830
- [Background] Lerman C, Schwartz M. Adherence and psychological adjustment among women at high risk for breast cancer. Breast Cancer Res Treat. 1993 Nov;28(2):145-55. doi: 10.1007/BF00666427. PMID 8173067